CLINICAL TRIAL: NCT02728544
Title: Post Exercise Irisin Levels in PWS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Prof. V. Gross, neuropediateic, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: shaaraZMC
Record Dates: First submitted 2016-02-17; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Prader Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Exercise; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prader Willi syndrome (Experimental): 16 (8 males) PWS adolescents and young adults
  Interventions: Other: exercise and blood tests
- Obese controls (Active Comparator): 16 - sex, age, and BMI-matched controls
  Interventions: Other: exercise and blood tests

INTERVENTIONS:
Other: exercise and blood tests — At an initial one-hour meeting study participants will learn to perform aerobic (treadmill) exercise and resistance training under the supervision of an experienced exercise physiologist. Exercise intensity will be assessed by direct measurement of VO2 m

SUMMARY:
Post exercise irisin levels in PWS patients Obesity, short stature, hypogonadism, hypotonia and impaired cognition are the major clinical features of Prader-Willi syndrome (PWS), a complex neurogenetic disorder due to lack of expression of paternal genes in the chromosomal region 15q11-13. Abnormal body composition with decreased muscle mass and increased fat mass contributes to low resting energy expenditure in PWS. Severe caloric restriction in the range of 800 kcal per day along with daily exercise regimens are needed to prevent weight gain and complications of obesity in this population.

Brown adipose tissue (BAT) once thought to be present only in infants, but now known to be present in adults as well, differs from the more abundant white adipose tissue (WAT) by dissipating energy through thermogenesis as a result of increased activity of the mitochondrial uncoupling protein (UCP-1). Recently evidence shows that exercise activates mitochondrial UCP-1 in subcutaneous WAT cells resulting in conversion of WAT to BAT-like adipocytes (Beige or BRITE adipose tissue). Various factors including natriuretic peptides, interleukin-6 and myokines (irisin, fibroblast growth factor 21, and ß-aminoisobutyric acid) appear to mediate the effects of exercising muscle on subcutaneous adipocytes.

Decreased amount and/or activity of BAT might contribute to the lower energy expenditure and extreme difficulty in weight-control in PWS. Lower levels or decreased myokine production could result in failure to convert subcutaneous WAT to Beige or BAT-like adipocytes, and therefore minimize or negate the otherwise beneficial metabolic effects of exercise. Direct measurement of peak oxygen uptake in PWS adults show that this population has markedly lower VO2 values compared with normal BMI-matched controls. BAT activity in vivo can be accurately measured only by performing PET/CT scans which include administrating radioactive tracers. For ethical reasons, direct assessment of BAT is not possible for purposes of clinical research in PWS individuals.

The investigators propose to study humoral responses to exercise in 16 (8 males) PWS adolescents and young adults and compare results with responses in a similar number of sex, age, and BMI-matched controls. At an initial one-hour meeting study participants will learn to perform aerobic (treadmill) exercise and resistance training under the supervision of an experienced exercise physiologist. Exercise intensity will be assessed by direct measurement of VO2 max. On a different day, a blood sample will be drawn before and immediately at the conclusion of the same exercise regimen. Blood samples will be assayed for irisin, interleukin-6, atrial natriuretic peptide, FGF-21, in addition to glucose, growth hormone, cortisol, norepinephrine, and lactate.

The investigators hypothesize that PWS participants will show weaker humoral responses to similar exercise regimens compared to normal control subjects. Data showing lower levels of myokines, such as irisin, following exercise in PWS might suggest that inadequate conversion of WAT to BAT-like adipocytes in subcutaneous adipose tissue results in decreased thermogenesis and abnormally low energy expenditure in this population. Potentially, development of pharmacologic agents which mimic irisin or other myokines by activating UCP-1 and converting WAT to BAT-like adipocytes could offer a new approach to weight-control in PWS individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult with Prader Willi syndrome

Exclusion Criteria:

* Inability to safely complete exercise regiment, heart disease or lungs disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal hormonal response | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gross Tsur Varda, Prof., Principal Investigator — Shaare Zedek Medical Center

IPD SHARING:
Plan to Share IPD: No